CLINICAL TRIAL: NCT01855022
Title: A Hospital-based Intervention Using Motivational Interviewing and Interactive Voice Response to Reduce Readmissions in Congestive Heart Failure and Chronic Obstructive Pulmonary Disease Patients: A Randomized Controlled Trial
Brief Title: A Trial to Reduce Readmissions Using Motivational Interviewing and Interactive Voice Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asante Health System (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ariel Linden, DrPH, President, Linden Consulting Group, LLC, Asante Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2AIT16621-B
Record Dates: First submitted 2013-05-10; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Congestive Heart Failure (CHF); Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Motivational interviewing; Interactive voice response; Hospital readmission
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MI + IVR (Experimental): 90 days of motivational interviewing and 30 days of interactive voice response monitoring
  Interventions: Behavioral: MI + IVR
- Usual Care (No Intervention): Usual care that a patient would receive absent the intervention

INTERVENTIONS:
Behavioral: MI + IVR — Participants in the intervention group received motivational interviewing from a registered nurse who is trained and proficient in this behavioral change modality. In addition, participants were instructed to make a daily toll-free call to an automated interactive voice response (IVR) system provided by Pharos Innovations® (Chicago, IL) for 30 days after discharge from the index admission. On each call patients heard a pre-recorded voice that goes through a series of questions about symptoms and the patient's daily weight. Information from the IVR system was automatically downloaded to a secure Internet site for review by the nurse at each hospital location.
  Arms: MI + IVR

SUMMARY:
The primary purpose of this study is to determine the effectiveness of a hospital-based intervention, using motivational interviewing and interactive voice response (IVR), to reduce hospital readmissions within 90 days of enrollment compared to usual care, for patients with heart failure and chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Recruitment and Enrollment of Participants:

Consented participants who met the criteria for either CHF or COPD, as identified via the daily hospital census report and using codes from the International Classification of Diseases, 9th Revision were randomized to either the treatment or control group. Participants who had mental or physical impairments that would prevent them from using the interactive voice response (IVR) system or communicating with the health coach were excluded. A study health coach visited the participant in their hospital room and, after explaining the study protocol, asked if they would like to participate and then consented them into the study if appropriate. After the participant signed the written consent, the health coach provided all participants with the 13-question set from the PAM and recorded the data. Lastly, the health coach assigned the study participant into either the treatment or control group using a pre-determined randomization system.

Description of the Intervention:

Control Group Activities:

Study staff did not interact with control group participants beyond the consenting and collection of PAM data, with the health coaches only interacting at baseline. Usual care occurred in the form of typical discharge planning by hospital staff, which consisted of providing brief traditional patient education before the participant was discharged.

Treatment Group Activities:

The intervention for the treatment group consisted of three components - Interactive Voice response (IVR), MI-based health coaching, and notification to the PCP.

First, participants used an interactive, voice telephony and web-based database system to monitor and improve their self-care behaviors and clinical status in the 30 days post discharge. Program participants were given the call-in number and followed through their first interaction with the system while they were still in the hospital, thereby ensuring their proficiency in the IVR functionality after discharge. Daily thereafter, participants were instructed to call in to the Tel-Assurance system using their cell phone, land-line, or via the internet. Participants entered into the Tel-Assurance system using a touch-tone phone or web browser and answered a set of daily survey questions that are customized to assess worsening of symptoms of their chronic disease. Information from the IVR system was automatically downloaded to a secure Internet site for review by the health coaches. The data was checked frequently and was displayed in such a way that participants' with "variances" were displayed at the top of the screen, flagging the coach's attention. Participants who triggered an alert for symptoms or out-of-range biometric values (such as increased body weight for congestive heart failure [CHF], or low forced expiratory volume for chronic obstructive pulmonary disease [COPD]), received a "same-day" follow-up call from the program health coach (who is also a registered nurse). If participants missed a daily call, they received an automated reminder call from the IVR service to encourage adherence. The health coaches also monitored adherence to the system and would call a participant if s/he had missed more than one day. Participants in the study were instructed that the IVR system was not to be used for urgent/emergent matters. They were also encouraged to call their health coach to discuss their symptoms or condition.

Second, participants received motivational interviewing (MI)-based health coaching, commencing while they are still in the hospital prior to discharge and for 90-days post-discharge. Motivational interviewing is a collaborative goal-oriented style of communication with particular attention to the language of change. It is designed to strengthen personal motivation of and commitment to a specific goal by eliciting and exploring the person's own reason for change within an atmosphere of acceptance and compassion. MI is an evidence-based patient-centered approach with four main principles: partnership, acceptance, compassion and evocation. There is a health coaching framework that provides structure for a provider to assist in being time-efficient in the coaching session: engaging, focusing, evoking, planning. In a review of literature of health coaching approaches, MI was found to be the only health coaching technique to be fully described and consistently demonstrated as causally and independently associated with positive behavioral outcomes. Health coaches received rigorous training in the MI approach and regular monitoring. Another optimal feature of MI is that there are validated standardized tools that have been developed to assess the fidelity of the provider/patient session to the approach. The Motivational Interviewing Treatment Integrity (MITI) tool was used during the training and active phases of the study to ensure that the coaches had achieved/maintained the level of proficiency that has been linked to clinical outcomes. Starting the health coaching process while the participant was still in the hospital was an attempt to ease the transition to the home by helping the participant understand the treatment plan and empower him/her to communicate in case there was a shift in health status that could result in a readmission. Continued health coaching sessions with the participant throughout the 90-day study period were provided to address the participant's activation level and, thus, the ability to self-manage his/her condition better. This approach was individually tailored to each participant based on their initial PAM score. In addition, the health coach discussed typical challenges with participants that they may face when recuperating from the hospital stay, such as understanding and following their treatment plan. Lastly, participants were empowered to take an active role in managing their condition and health, including appropriate and timely interaction with their PCP when a problem arose that could lead to a deterioration of their health status. If the participant was readmitted to the hospital during the study period, the health coach provided follow up with the participant and the PCP to determine the best course of action. In addition, study staff determined the cause of the readmission and recorded it for analysis, which was performed and discussed by study staff on an on-going basis throughout the study period.

Third, the investigators attempted to engage the participant's primary care provider (PCP) in the care plan by directly providing them with the discharge summary upon the participant's release from the hospital. Informing the PCP of the participant's hospitalization should have increased the likelihood the PCP's office would be proactive in reaching out to the participant to schedule a follow-up office visit. The provider was encouraged to: (a) schedule an office visit with the participant; and (b) to communicate directly with the health coach to suggest areas of focus for the care plan. The investigators were not successful in getting any of the PCP's to contact the health coaches to discuss their patient's progress or health plans.

Outcome Measures:

All outcomes were analyzed separately for each of the two conditions, congestive heart failure (CHF) and chronic obstructive pulmonary disease (COPD). The investigators' primary outcomes for this study were readmissions, hospital days, and emergency department visits occurring within 90 days of discharge from the index admission. The investigators' secondary outcomes were 90 day mortality and patient activation measure scores at 30 and 90 days. The investigators further review statistics relating to the IVR technology used to track treatment patients' disease specific symptoms. All analyses were conducted using the intention to treat approach.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Index hospitalization for congestive heart failure or chronic obstructive pulmonary disease
* Access to telephone

Exclusion Criteria:

* Cognitive impairment
* Resident of a nursing home
* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Hospital readmission rate (all cause) | 90 days
  Readmissions within 90 days from discharge of the index admission, for any diagnosis

SECONDARY OUTCOMES:
Emergency department visit rate (all cause) | 90 days
  Visits to the emergency department within 90 days from discharge of the index admission, for any diagnosis
Hospital days (all cause) | 90 days
  The total number of hospitals days for those readmissions occurring in the 90 day period after discharge of the index admission
Mortality | 90 days
  Deaths occurring within 90 days of discharge of the index admission
Patient Activation Measure (PAM) score | 90 days
  Patient Activation Measure (PAM) score at 30 and 90 days post discharge of the index admission

OTHER OUTCOMES:
Days compliant with interactive voice response system (treatment group only) | 30 days
  The average number of days that treatment group participants engaged with the interactive voice response system

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Linden, DrPH, Principal Investigator — Linden Consulting Group, LLC; Debra Flickinger, BS, Study Director — Asante Health System
Locations (2):
- United States (2):
  - Asante Three Rivers Medical Center, Grants Pass, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon

REFERENCES:
- [Derived] Linden A, Butterworth S. A comprehensive hospital-based intervention to reduce readmissions for chronically ill patients: a randomized controlled trial. Am J Manag Care. 2014 Oct;20(10):783-92. PMID 25365681